CLINICAL TRIAL: NCT01711788
Title: A New Approach to Improve Long-term Hematopoietic Recovery After Allogeneic Umbilical Cord Blood Transplantation in Children - Intrabone Infusion of Umbilical Cord Blood Stem Cells
Brief Title: Intrabone Infusion of Umbilical Cord Blood Stem Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henrique Bittencourt, MD, PhD (Other)
Collaborators: Michel Duval, MD (Unknown); Pierre Teira, MD (Unknown); Sonia Cellot, MD, PhD (Unknown); Isabelle Louis, PhD (Unknown); Elie Haddad, MD, PhD (Unknown); Marie-France Vachon, MScN (Unknown); Marion Cortier, PhD (Unknown)
Responsible Party: Sponsor-Investigator, Henrique Bittencourt, MD, PhD, Hematologist - Oncologist, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB-UCBT
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Hematopoietic stem cells; Umbilical cord blood transplantation; Intrabone infusion; Platelet recovery; Neutrophil recovery; Pediatric patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intrabone umbilical cord blood tranplant (Experimental): Intrabone infusion of umbilical cord blood stem cells
  Interventions: Procedure: Intrabone infusion of umbilical cord blood stem cells

INTERVENTIONS:
Procedure: Intrabone infusion of umbilical cord blood stem cells

SUMMARY:
The purpose of this study is to determine if the method of intrabone infusion of hematologic stem cells can increase and accelerate hematopoietic reconstitution after umbilical cord blood transplantation in pediatric patients.

DETAILED DESCRIPTION:
Umbilical cord blood transplantation (UCBT) has been increasingly used to treat malignant and non-malignant haematological, immunodeficiency and some metabolic diseases. UCBT offers the advantages of easy procurement, no risk to donors, a reduced risk of transmitting infections, immediate availability of cryopreserved units, and acceptable partial HLA mismatches. However, patients treated with UCBT show delayed hematopoietic and immunological recoveries, have higher rates of infection, and relapse from the original malignant disease, which can all lead to life threatening problems. UCBT can also result in a higher rate of graft failure compared to other hematopoietic stem cell transplantation (HSCT) sources. The problem of a slower hematopoietic recovery post-UCBT has been addressed using a number of different approaches in adult patients.In adults, use of intrabone injection of cord blood results in a faster hematopoietic recovery in a phase II study. However, there is no clinical trial in pediatric patients.

This study is addressed to determine if a change in the cord blood stem cell infusion method can increase and accelerate hematopoietic reconstitution after UCBT in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* One to 21 years of age;
* More than 10 kg in weight;
* Diagnosis of hematopoietic disorders (malignant or not) with an indication for hematopoietic stem cell transplantation;
* Absence of an HLA-identical related donor;
* Availability of a single cord blood (CB) with at least 3 x 10^7 nucleated cells (NCs)/kg (if HLA identical or 1 HLA-mismatch) or at least 4 x 10^7 NCs/kg (if a 2 HLA-mismatch) at freezing. Use of two CB units ("double cord transplant") will be allowed provided that: 1) a single CB unit fulfilling the above criteria is not available; 2) a maximum of 2 HLA mismatch is present for each CB unit; and 3) a minimum of 4 x 10^7 NCs/kg (as the sum for both CB units) is present at freezing.
* A myeloablative-conditioning regimen;
* A Lansky (for patients less than 16 years of age) or Karnofsky (for patients more than 16 years of age) score equal to or higher than 70%.
* Adequate organ function as follows:
* Cardiac (ejection fraction > 50%);
* Renal (serum creatinine within the normal range for age, and creatinine clearance or a GFR > 70 ml/min/1.73m2);
* Hepatic (AST or ALT < 5 x upper limit of normal for age);
* Pulmonary (FEV1, FVC, and DLCO ≥ 50% by pulmonary function tests or, in children unable to cooperate, no sign of dyspnea at rest, no exercise intolerance, no supplementary oxygen therapy, and a normal pulmonary radiography or pulmonary scan);
* No sign of uncontrolled systemic bacterial, fungal or viral infection;
* Written informed consent by the patient or his/her legal guardian

Exclusion Criteria:

* Non-myeloablative conditioning;
* Pregnancy or breastfeeding;
* HIV positive serology;
* Bone disease (e.g. osteopetrosis, osteogenesis imperfecta)
* Previous autologous or allogeneic hematopoietic stem cell transplantation performed up to one year before enrolment, except in the case of non-engraftment or early rejection of a previous allogeneic stem cell transplantation.
* Active skin infection at the site of intrabone injection.
* History of intolerance/allergy to sedation medications or local anesthetics.
* Contraindication to sedation

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Platelet recovery rate | at 100 days post- transplantation
  First of seven days of untransfused platelet count higher than 20 x 10^9/L

SECONDARY OUTCOMES:
Neutrophil recovery rate | at 60 days post- transplantation
  First of three days of absolute neutrophil count equal or higher than 0.5 x 10^9/L
Immunological reconstitution | at 30, 60, 100, 180, and 360 days post- transplantation
  Total number of T cells (and subpopulations), B and NK (natural killer) cells in peripheral blood at different time-points
Donor chimerism rate | at 30, 60,100, and 180 days post-transplantation
  Percentage of donor(s) cells in peripheral blood at different time-points
Acute GVHD (grade 2-4) rate | at 180 days
  Incidence of grade II-IV acute GVHD (Graft versus Host Disease)
Infection rate (bacterial, viral, fungal and parasitic) | at 180 days post-transplantation
  Clinical and microbiological documented infections will be reported according to anatomic site, date of onset and microorganism
Event-free and overall survival | at 2 years
  Event-free survival is defined as the time interval between transplantation and relapse, graft rejection, death or last follow-up, whichever occurs first; Overall survival is defined as the time between transplantation and death or last follow-up
Adverse infections (grade and frequency) | at one month post-transplantation
  Toxicity will be assessed using the Common Terminology Criteria for Adverse Events v4.0
chronic GVHD | at 2 years post-transplantation
  Incidence of chronic GVHD (Graft versus Host Disease) will be scored according to NIH consensus on chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Henrique Bittencourt, MD, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Vairy S, Louis I, Vachon MF, Richer J, Teira P, Cellot S, Villeneuve E, Haddad E, Duval M, Bittencourt H. Intrabone infusion for allogeneic umbilical cord blood transplantation in children. Bone Marrow Transplant. 2021 Aug;56(8):1937-1943. doi: 10.1038/s41409-021-01275-0. Epub 2021 Apr 6. PMID 33824433